CLINICAL TRIAL: NCT02387671
Title: Evaluation of mHealth Counseling for Lifestyle Behaviors Among Breast Cancer Survivors
Brief Title: Weight Management Among Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Boston University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-33650
Record Dates: First submitted 2015-02-12; First posted 2015-03-13 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2015-01

CONDITIONS: Body Weight
MeSH Terms: conditions — Body Weight | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mHealth Platform (Experimental): The primary interventions employed in the study are wifi enabled tracking devices, text message communications and behavioral counseling.
  Interventions: Behavioral: Device: FitBit Flex wrist band; Behavioral: Device: FitBit Aria weight scale; Behavioral: Diet Intake Messages; Behavioral: Behavioral Counseling

INTERVENTIONS:
Behavioral: Device: FitBit Flex wrist band — Participants will track their daily steps walked and hours of sleep by wearing the FitBit Flex wrist band during the 8 week study period. The data collected from the wrist band will be synced to participants' FitBit smart phone application and monitored by the study team.
  Other Names: FitBit Flex™
Behavioral: Device: FitBit Aria weight scale — Participants will record their daily body weight during the 8 week study period by stepping on the FitBit Aria weight scale. The data collected from the scale will be synced to participants' FitBit smart phone application accounts and monitored by the study team.
  Other Names: FitBit Aria® wi-fi smart scale
Behavioral: Diet Intake Messages — The study team will send participants daily text messages regarding their dietary intake. Each message will contain five questions that yield a yes, or no response. Messages will be sent daily during the 8 week study period. Responses from the messages will be recorded and monitored by the study team to enhance the behavioral counseling intervention.
Behavioral: Behavioral Counseling — Participants will engage in four phone calls with the study counselor to discuss behavioral several topics (physical activity, sleep, fatigue & dietary patterns) and to reflect on their data recorded by the FitBit devices. The calls will take place on a bi-weekly basis. During the weeks between calls, the counselor will maintain contact with the participants through asynchronous text messages to monitor their progress in the study.

SUMMARY:
The long-term goal of this research is to develop, evaluate and implement effective mHealth technology interventions that improve cancer management outcomes by changing lifestyle behaviors among urban health- disparity facing populations. To accomplish this goal, the investigators will need to determine the feasibility and preliminary efficacy of an intervention in which breast cancer survivors receive counseling about lifestyle behaviors (weight, nutrition, and physical activity) from a health counselor trained in evidenced-based behavioral counseling methods.

DETAILED DESCRIPTION:
Tremendous advances in detection and treatment of breast cancer have led to an increasingly large cohort of survivors focused on health promotion and reducing the risk of recurrence. While adjuvant therapy, such as hormone therapy, is often used to prevent cancer recurrence, modification of lifestyle is an effective tool to increase quality of life, prevent future cancer recurrence and increase long-term health. However, translating these recommendations into population-wide, inexpensive, sustainable programs for cancer survivors has to date proven largely unrealized. These programs are particularly needed in health disparity-facing populations (i.e., low socio-economic status and/or racial/ethnic minority groups) due to the high burden of cancer incidence and mortality they face. Limited translation is due to many factors including the complexity of lifestyle habits, high patient burden of many behavioral interventions, low levels of engagement and adherence to interventions, and the lack of integration of behavior change tools into daily lifestyles. In this context, there is great promise of tools that are mobile, simple, and embedded into daily life routines. The long-term goal of this research program is to develop, evaluate and implement effective mHealth technology interventions that improve cancer management outcomes by changing lifestyle behaviors among urban health- disparity facing populations.

The mHealth intervention for cancer survivors devised by the investigators consists of several components: 1) a commercially available smart phone app that captures patients' behavioral data (steps, sleep, weight) using devices (a FitBit and a FitBit scale), 2) text messages to participants to collect additional data (foods eaten, eating habits), and 3) phone sessions with a non-professionally trained health counselor about diet and physical activity behaviors.

The investigators propose to test the feasibility and preliminary outcomes on weight, behaviors, psychological factors as well as participant engagement in the intervention of our mHealth counseling intervention among 20 breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in intervention by sharing FitBit account information (log in/password) with study team
* 6 months or more since receiving cancer treatment including surgery, radiation, or chemotherapy (self-reported)
* 2 or more years post breast cancer diagnosis (self-reported)
* Current ownership of an iOS or Android based platform smartphone and home wifi
* Age 18 and above
* Ability to speak and read in English
* Overweight or obese (body mass index ≥ 25)
* Female

Exclusion Criteria:

* Medical conditions including dementia, active cancer, anorexia or any other condition in the opinion of the investigator makes the participant unsuitable for inclusion in the study
* Presence of a pacemaker or other internal medical device
* Those with contraindications for physical activity
* Pregnant women
* Inability to easily navigate programs on a smartphone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Body Weight | 8 weeks
  Participants will register daily body weight measurements during the 8-week study period. Weight will be recorded in units of pounds using the FitBit wifi compatable. All data will be synced to the participants' FitBit account and monitored by the study team.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Quintiliani, Ph.D., Principal Investigator — Assistant Professor
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Quintiliani LM, Mann DM, Puputti M, Quinn E, Bowen DJ. Pilot and Feasibility Test of a Mobile Health-Supported Behavioral Counseling Intervention for Weight Management Among Breast Cancer Survivors. JMIR Cancer. 2016 Jan-Jun;2(1):e4. doi: 10.2196/cancer.5305. Epub 2016 May 9. PMID 27761518